CLINICAL TRIAL: NCT05578495
Title: Association of a Digital Signature of Physical Activity and Sedentary Lifestyle With the Development of Multimorbidities Over 4 Years of Follow-up in Chronic Diseases (eMOB) : a Prospective Cohort
Brief Title: Association of a Digital Signature of Physical Activity and Sedentary Lifestyle With the Development of Multimorbidities in Chronic Diseases (eMOB)
Acronym: eMOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2021 TOURNADRE; 2021-A01967-34 (Other: ANSM)
Record Dates: First submitted 2022-09-19; First posted 2022-10-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Exercise; Sedentary Behavior; Non Communicable Diseases; Comorbidities and Coexisting Conditions; Comorbidity; Multimorbidity; Digital Technology
Keywords: Physical Activity; Sedentary Lifestyle; Chronic Diseases; Comorbidities; Multimorbidity; Personal digital health; Personalized medecine
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Noncommunicable Diseases; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic diseases (Other): Cohort Study
  Interventions: Other: Accelerometer data

INTERVENTIONS:
Other: Accelerometer data — Patients will wear an accelerometer 3 times a year for 5 days (3 weekdays and 2 weekend days), the data will be collected

SUMMARY:
Physical activity (PA) and sedentary lifestyle are determinants in the development of chronic diseases and associated quality of life alterations. PA levels are correlated with quality of life and morbidity in chronic lung disease (COPD), cardiovascular disease, diabetes, cancer, chronic inflammatory rheumatism, fibromyalgia and anxiety disorders. In these diseases, low-intensity PA often represents the main PA and the quantity of PA is correlated with health parameters.

This study aims to identify a typical profile (signature) in relation to the appearance of other chronic diseases, complications of your disease, from recording your physical activity and sedentary lifestyle by sensors evaluating very precisely the movements and taking into account the characteristics and disability related to your disease. The results of this study would therefore make it possible to identify this signature even before the appearance of complications or other diseases.

DETAILED DESCRIPTION:
Study design :

eMOB study is a monocentric prospective cohort study. We aim to explore in a longitudinal study the association of a digital signature of PA and sedentary lifestyle with the development of at least one additionnal comorbidity overs 4 years of follow-up in chronic diseases.

Population :

Patients with inflammatory rheumatic disease(rheumatoid arthritis and spondyloarthritis), pre-surgical knee and hip osteoarthritis, major depressive disorder and bipolar disorder, type 2 diabetes, obesity, COPD and chronic pain followed up in the observational cohorts specific to each pathology at the CHU of Clermont Ferrand, will be proposed to participate in the study during their follow-up visit.

Method :

The occurrence of comorbidity is monitored every year during follow-up visits of the patients. Physical activity and sedentary lifestyle is assessed using accelerometer and wearable sensors. The combination of quantitative analysis of movement with a more detailed analysis of movement and sequences of movements, and a personalization of the algorithm according to the disease and the context, could make it possible to establish predictive signatures either of the disease itself or of associated complications.

700 patients will be included in the study.They will be followed for 4 years with :

* An annual visit during which :

  * clinical data in the routine follow-up will be collected (BMI, waist circumference, blood pressure, heart rate, comorbidities, activity and severity scores specific to each disease and used for the routine follow-up, treatments, lifestyle, family and socio-professional situation, education level)
  * comorbidities will be noted by the list used for the study
  * physical capacity will be assessed with the 6-minute walk test and the hand grip
  * questionnaires about Pain (QCD), Fatigue (FACIT-F), Anxiety and Depression (HADs), Quality of life (WhoQol-BREF), Poverty (EPICES), Physical activity questionnaire (RPAQ), Barriers and Facilitators to physical activity questionnaire (B&F-AP), Sleep and daytime sleepiness (PSQI and Epworth), treatment compliance (MARS) will be completed
  * specific data for each pathology in each cohort will be collected
* Accelerometer data 3 times a year for 5 days (3 weekdays and 2 weekend days) will be collected
* Electronic patient report outcomes (e-PRO) every 4 months concerning the socio-professional situation of the patients, alcohol and tobacco consumption, skipping meals and snacking between meals, health problems they may encounter during the study. Numerical scales between 0 and 10 will be completed to assess disease status, health status, pain, sleep, fatigue, psychological well-being, and anxiety.

Among the included patients, 10 patients per cohort will participate in the preliminary feasibility phase of the study before starting the follow-up in the study. It is a validation of the acquisition modalities of the pre-selected sensors and a calibration on representative samples of patients with the different chronic pathologies studied (locomotor, respiratory, metabolic, psychiatric, pain).

ELIGIBILITY:
Inclusion Criteria:

* Patient follow-up at CHU Clermont-Ferrand for a chronic disease in one of the following observational cohorts:

  * Inflammatory rheumatic disease(rheumatoid arthritis, spondyloarthritis) included in the RCVRIC cohort (CPP Sud-Est VI N° ID-RCB- A01847-40)
  * Pre-surgical knee and hip osteoarthritis (Evalmob) (ID-RCB N° 2019- A01017-50)
  * Major depressive disorder included in the FACE-DR cohort (CNIL agreement: DR- 2015-673) and Bipolar disorder included in the FACE-BD cohort (CPP Ile de France IX; January 18, 2010) of the Adult Psychiatry Department B
  * Type 2 diabetes included in the cohort of the sport medicine service "Rehabilitation T2" (CNIL agreement 0164)
  * Obesity included in the "Obesity" sports medicine service cohort (CNIL agreement 0164)
  * COPD included in the "COPD Rehabilitation" sports medicine service cohort (CNIL agreement 0164)
  * Chronic pain cohort (eDOL) (CPP West II N° ID-RCB 2020-A02027-32)
* Affiliation to a social security system.
* Able to provide written informed consent to participate in the research.

Exclusion Criteria:

* Inability to practice physical activity
* Pregnant or breastfeeding
* Refusal to participate
* Minors or adults under the protection of the law or under the protection of justice.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of one additional comorbidity in patients with chronic diseases. | year 4
  Association of a digital signature of PA and sedentary lifestyle with the development of at least one additional comorbidity over 4 years of follow-up.
Digital signature of sedentary lifestyle and PA in patients with chronic diseases. | Year 4
  A sensor of movement will be worn by the patients for 5 days every 4 months during the study, to detect and quantify the physical activity and the sedentarity according to their intensity. This sensor will be accelerometer, allowing the acquisition of movements second by second. The analysis of the data from the sensors, the occurrence of a new comorbidity, the clinical data will allow to establish an algorithm to define a profile (digital signature) of occurrence of a new chronic disease.

SECONDARY OUTCOMES:
Occurence of multimorbidity in patients with chronic diseases. | Year 1
  Association of a sedentary and PA signature with the development over 4 years of one, two, three, or more comorbidities (multimorbidity).
Occurence of multimorbidity in patients with chronic diseases. | year 2
  Association of a sedentary and PA signature with the development over 4 years of one, two, three, or more comorbidities (multimorbidity).
Occurence of multimorbidity in patients with chronic diseases. | Year 3
  Association of a sedentary and PA signature with the development over 4 years of one, two, three, or more comorbidities (multimorbidity).
Occurence of multimorbidity in patients with chronic diseases. | Yaer 4
  Association of a sedentary and PA signature with the development over 4 years of one, two, three, or more comorbidities (multimorbidity).
Correlation of PA/sedentary signature with destabilization or improvement/stability of the chronic condition. | Year 1
  Collect during the study clinical data, disease activity parameters in each cohort, physical capacity, and self questionnaires to explore PA/sedentary signature and its trajectory associated with destabilization or improvement/stability of the chronic condition.
Correlation of PA/sedentary signature with destabilization or improvement/stability of the chronic condition. | Year 2
  Collect during the study clinical data, disease activity parameters in each cohort, physical capacity, and self questionnaires to explore PA/sedentary signature and its trajectory associated with destabilization or improvement/stability of the chronic condition.
Correlation of PA/sedentary signature with destabilization or improvement/stability of the chronic condition. | Year 3
  Collect during the study clinical data, disease activity parameters in each cohort, physical capacity, and self questionnaires to explore PA/sedentary signature and its trajectory associated with destabilization or improvement/stability of the chronic condition.
Correlation of PA/sedentary signature with destabilization or improvement/stability of the chronic condition. | Year 4
  Collect during the study clinical data, disease activity parameters in each cohort, physical capacity, and self questionnaires to explore PA/sedentary signature and its trajectory associated with destabilization or improvement/stability of the chronic condition.
Correlation of PA/sendetary and treatments for chronic diseases. | Year 1
  Collect treatments of patients in each cohort at inclusion and each year over the study to explore PA/sedentary signature and its trajectory associated with achieving a decline in background treatments for chronic disease.
Correlation of PA/sendetary and treatments for chronic diseases. | year 2
  Collect treatments of patients in each cohort at inclusion and each year over the study to explore PA/sedentary signature and its trajectory associated with achieving a decline in background treatments for chronic disease.
Correlation of PA/sendetary and treatments for chronic diseases. | Year 3
  Collect treatments of patients in each cohort at inclusion and each year over the study to explore PA/sedentary signature and its trajectory associated with achieving a decline in background treatments for chronic disease.
Correlation of PA/sendetary and treatments for chronic diseases. | Year 4
  Collect treatments of patients in each cohort at inclusion and each year over the study to explore PA/sedentary signature and its trajectory associated with achieving a decline in background treatments for chronic disease.
Correlation of PA and sedentary measures and quality of life (QOL) of patients | Year 1
  Quality of life will be assessed with the World Health Organization Quality of Life Instruments (WhoQol-BREF) questionnaire, which has 26 items, divided into 4 domains: physical health, psychological, social relationship and environment. The score for each item ranges from 1 to 5. The score for each domain is calculated using a template designed by the WhoQol-BREF development team. The higher the score, the better the health status.
  The association between the score of each domain of WhoQol-BREF and PA/sedentary profile will be explored.
Correlation of PA and sedentary measures and quality of life (QOL) of patients | Year 2
  Quality of life will be assessed with the World Health Organization Quality of Life Instruments (WhoQol-BREF) questionnaire, which has 26 items, divided into 4 domains: physical health, psychological, social relationship and environment. The score for each item ranges from 1 to 5. The score for each domain is calculated using a template designed by the WhoQol-BREF development team. The higher the score, the better the health status.
  The association between the score of each domain of WhoQol-BREF and PA/sedentary profile will be explored.
Correlation of PA and sedentary measures and quality of life (QOL) of patients | year 3
  Quality of life will be assessed with the World Health Organization Quality of Life Instruments (WhoQol-BREF) questionnaire, which has 26 items, divided into 4 domains: physical health, psychological, social relationship and environment. The score for each item ranges from 1 to 5. The score for each domain is calculated using a template designed by the WhoQol-BREF development team. The higher the score, the better the health status.
  The association between the score of each domain of WhoQol-BREF and PA/sedentary profile will be explored.
Correlation of PA and sedentary measures and quality of life (QOL) of patients | Year 4
  Quality of life will be assessed with the World Health Organization Quality of Life Instruments (WhoQol-BREF) questionnaire, which has 26 items, divided into 4 domains: physical health, psychological, social relationship and environment. The score for each item ranges from 1 to 5. The score for each domain is calculated using a template designed by the WhoQol-BREF development team. The higher the score, the better the health status.
  The association between the score of each domain of WhoQol-BREF and PA/sedentary profile will be explored.
Occurrence of hospitalization and/or surgery of patients in each cohort | Year 1
  Patient hospitalization and/or surgery data are collected during follow-up (period of hospitalization, condition of hospitalization).
Occurrence of hospitalization and/or surgery of patients in each cohort | Year 2
  Patient hospitalization and/or surgery data are collected during follow-up (period of hospitalization, condition of hospitalization).
Occurrence of hospitalization and/or surgery of patients in each cohort | Year 3
  Patient hospitalization and/or surgery data are collected during follow-up (period of hospitalization, condition of hospitalization).
Occurrence of hospitalization and/or surgery of patients in each cohort | Year 4
  Patient hospitalization and/or surgery data are collected during follow-up (period of hospitalization, condition of hospitalization).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Tournadre, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France